CLINICAL TRIAL: NCT03178019
Title: Dipeptidyl Peptidase 4 (DPP4) Activity and Its Associations With Endothelial Dysfunction, Inflammatory and Metabolic Markers, Heart Rate and Blood Pressure Variability, and Measures of Adiposity in Subjects With Different Grades of Glucose Tolerance
Brief Title: DPP4 Activity, Microvascular Reactivity and Inflammation
Acronym: DPP4
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Professor, Rio de Janeiro State University
Other Study IDs: 940.029
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Overweight; Pre Diabetes; Diabetes Mellitus Type 2 Without Complication
MeSH Terms: conditions — Overweight; Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Euglycemia group: Normoglycemic/normotolerant subjects
  Interventions: Other: Laser-Doppler methods
- Prediabetes group: Subjects with prediabetes
  Interventions: Other: Laser-Doppler methods
- Diabetes group: Subjects with type 2 diabetes mellitus
  Interventions: Other: Laser-Doppler methods

INTERVENTIONS:
Other: Laser-Doppler methods — This was a cross-sectional study in which participants were subjected to a screening phase before being eligible to participate in the study. All subjects were submitted to Laser-Doppler methods (assessment of microcirculatory blood flow), bioimpedance analysis (assessment of body composition), venous blood collections (laboratory analysis), and Finometer Pro (assessment of heart rate variability and blood pressure variability).
  Other Names: Venous blood collections; Bioimpedance analysis; Finometer Pro

SUMMARY:
Dipeptidyl peptidase 4 (DPP4) is a serine exopeptidase able to inactivate various oligopeptides involved in inflammation, immunity and vascular function. Our aim was to investigate the associations between constitutive levels of DPP4 activity and inflammatory biomarkers, skin microvascular reactivity, gut peptides, insulin resistance indexes, heart rate and blood pressure variability, and measures of adiposity in subjects with different grades of glucose tolerance.

DETAILED DESCRIPTION:
Dipeptidyl peptidase 4 (DPP4), also known as adenosine deaminase binding protein or cluster of differentiation 26 (CD26), is a serine exopeptidase able to inactivate various oligopeptides composed of proline, hydroxyproline, or alanine as the penultimate residue. In recent years, DPP4 has received attention due to its ability to rapidly inactivate the main incretins secreted by the gastrointestinal tract: glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP). As its own name already says, incretins enhance insulin secretion in a glucose-dependent fashion, but also suppress or modulate glucagon secretion. Since it was demonstrated that type 2 diabetes mellitus (T2D) have incretin deficiency and hyperglucagonemia on its physiopathology, gliptins emerged as a new class of drugs for the treatment of this disease, acting through the inhibition of DPP4 and consequently ameliorating these defects.

DPP4 not only inactivate incretins but also a number of cytokines, chemokines, and neuropeptides involved in inflammation, immunity and vascular function. Furthermore, evidence from in vitro and in vivo studies, including clinical ones in T2D, suggested that gliptins' inhibition of DPP4 was associated with reduction of inflammatory biomarkers and also attenuation of endothelial dysfunction and atherogenesis, possibly through regulation of the DPP4 substrates.

There is a paucity of studies that associate the constitutive levels of DPP4 activity (i.e., outside the context of pharmacological inhibition of the enzyme) with markers of inflammation and endothelial function, specially tested on skin microcirculation. We hypothesized that constitutive levels of DPP4 activity might be directly associated to inflammation and inversely correlated with skin blood flux and one or more components of vasomotion (suggesting an association with endothelial disfunction) even in the absence of diabetes. Our aim was to investigate the associations between constitutive levels of DPP4 activity and inflammatory biomarkers, skin microvascular reactivity, gut peptides, insulin resistance indexes, heart rate and blood pressure variability, and measures of adiposity in subjects with different grades of glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25.0 kg/m²
* Any degree of glucose tolerance

Exclusion Criteria:

* BMI < 25.0 kg/m²
* Uncontrolled chronic diseases, such as arterial hypertension
* Smoking
* Severe alcoholism
* Moderate to severe chronic kidney disease, heart failure, chronic lung disease, and chronic liver disease
* Fasting serum triglycerides > 400 mg/dl
* Fasting serum cholesterol > 300 mg/dl
* Pregnancy and breastfeeding
* Women in the climacteric period
* Individuals who undergo bariatric surgery
* Acute disease at the time of sampling
* Initiation of statin or change in its dose within 60 days
* Use of aspirin and/or fluconazole within 10 days prior to the exams

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men and women aged between 18 and 50 years, BMI ≥ 25.0 kg/m², with different degrees of glucose tolerance, and living in the state of Rio de Janeiro (Brazil).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Intergroup analysis of the associations between DPP4 activity and skin microvascular reactivity | 63 minutes
  Intergroup analysis of the associations between DPP4 activity and skin microvascular reactivity (blood flux and vasomotion evaluated by Laser-Doppler methods) - baseline assessment and at 30 and 60 min after a standardized meal intake (ingested over 3 minutes)
Intergroup analysis of the associations between DPP4 activity and markers of inflammation | 63 minutes
  Intergroup analysis of the associations between DPP4 activity and markers of inflammation - baseline assessment and at 30 and 60 min after a standardized meal intake (ingested over 3 minutes)

SECONDARY OUTCOMES:
Intergroup analysis of the associations between DPP4 activity and biochemical parameters | 63 minutes
  Intergroup comparisons between the associations of DPP4 activity and Biochemical parameters (including gut peptides) - baseline assessment and at 30 and 60 min after a standardized meal intake (ingested over 3 minutes)
Intergroup analysis of the associations between DPP4 activity and insulin resistance indexes, heart rate and blood pressure variability, and measures of adiposity | Baseline evaluation
  Intergroup analysis of the associations between DPP4 activity and insulin resistance indexes, heart rate and blood pressure variability (evaluated by Finometer Pro), and measures of adiposity at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wellington S Silva Júnior, MD, Principal Investigator — State University of Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No